CLINICAL TRIAL: NCT02122055
Title: Sequential Use of Propofol/Midazolam and Dexmedetomidine for Sedation in Mechenical Ventialtion Patients in ICU, A Randomized Controlled Study.
Brief Title: Sequential Use of Propofol/Midazolam and Dexmedetomidine for Sedation in Mechenical Ventialtion Patients in ICU.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMATJHICU
Record Dates: First submitted 2014-04-21; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Mechanical Ventilation Complication
Keywords: combined sedation
MeSH Terms: interventions — Fentanyl; Propofol; Midazolam; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol/Dexmedetomidine (Experimental): 1. Propofol is started with dosage of 0.3 mg/kg/h, observe the patient's response, increase 0.3 mg/kg/h propofol every 10 minutes until target sedation level is obtained(Riker Sedation Agitation Score(SAS) 3-4),then 0.3-3 mg/kg/h propofol is maintained.
  2. After the screen of the weaning is passed, change to Dexmedetomidine sedation, the dose is 0.2-0.7 mg/kg/h and continuously pumped, increase the dose 0.1-0.2 mg/kg/h every 30 minutes, titrate to Riker Sedation Agitation Score(SAS) 3-4，the maximum dose is 1 mg/kg/h maintained，and prepare for weaning.
  Interventions: Drug: Fentanyl; Procedure: Sedation assessment; Procedure: Screen of weaning; Drug: Propofol; Drug: Dexmedetomidine
- Midazolam/Dexmedetomidine (Experimental): 1. Midazolam 2 mg is slowly titrated to Riker Sedation Agitation Score(SAS) 3-4 every 10 minutes, then Midazolam 0.02-0.1 mg/kg/h is maintained.
  2. After the screen of the weaning is passed, change to Dexmedetomidine sedation, the dose is 0.2-0.7 mg/kg/h and continuously pumped, increase the dose 0.1-0.2 mg/kg/h every 30 minutes, titrate to Riker Sedation Agitation Score(SAS) 3-4，the maximum dose is 1 mg/kg/h maintained，and prepare for weaning.
  Interventions: Drug: Fentanyl; Procedure: Sedation assessment; Procedure: Screen of weaning; Drug: Midazolam; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 0.7-1μg/kg，prn pain assessment is done every 4 hours，maintain Behavioral Pain Scale（BPS） 0-2.
Procedure: Sedation assessment — Sedation assessment is done every 4 hours,maintain the Riker Sedation Agitation Score(SAS) 3-4.
Procedure: Screen of weaning — 1. Screen of weaning is done at 8:00 every morning. 2 If the patient is successful to wean, stop the Dexmedetomidine sedation. 3. If failed to wean, the patient is ventilated again and try to wean after 24 hours, until it is successful to wean and stop sedation，
Drug: Propofol — Propofol is started with dosage of 0.3 mg/kg/h, observe the patient's response, increase 0.3 mg/kg/h propofol every 10 minutes until target sedation level is obtained(Riker Sedation Agitation Score(SAS) 3-4),then 0.3-3 mg/kg/h propofol is maintained.
  Arms: Propofol/Dexmedetomidine
Drug: Midazolam — Midazolam 2 mg is slowly titrated to Riker Sedation Agitation Score(SAS) 3-4 every 10 minutes, then Midazolam 0.02-0.1 mg/kg/h is maintained.
  Other Names: Liyuexi
  Arms: Midazolam/Dexmedetomidine
Drug: Dexmedetomidine — After the screen of the weaning is passed, change to Dexmedetomidine sedation, the dose is 0.2-0.7 mg/kg/h and continuously pumped, increase the dose 0.1-0.2 mg/kg/h every 30 minutes, titrate to Riker Sedation Agitation Score(SAS) 3-4，the maximum dose is 1 mg/kg/h maintained，and prepare for weaning.
  Other Names: Yisi

SUMMARY:
For the patient who passed the screen of weaning from ventilation, the traditional sedation drug such as propofol and midazolam should be decreased or stopped, then it would induce the stress response and agitation, such as hypertension,tachycardia etc. In order to resolve that problem, the sedation should be given again. but if renewed to sedation, it would cause prolonged sedation and ventilation duration.

So as to resolve above issues, after the patient passed the screen of weaning, sedation is changed to Dexmedetomidine, a new sedation drug, that could wake up at any time. So our study to compare the efficacy and safety of sequential sedation of propofol or midazolam and dexmedetomidine in mechanical ventilated ICU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Anticipated Ventilation and sedation duration of at least 48 hours
3. Age≥18 years old
4. Weight is in the range of ±20% of standard weight.[Standard weight= (Height(cm)-80)×70﹪ for male and (Height(cm)-70)×60﹪for female] -

Exclusion Criteria:

1. Extremely unstable of circulatory system, such as systolic blood pressure less than 90 mm Hg despite continuous infusions of vasopressors before the start of study drug infusion or shock；
2. Heart rate less than 50 bpm
3. Second or third degree heart block
4. Serious central nervous system pathology(acute stroke, uncontrolled seizures,severe dementia)
5. Acute hepatitis or severe liver disease (Child-Pugh class C)
6. Dialysis of all types 7）History of neuromuscular disease

8) Unstable mental status and metal illness 9) Sure or suspected abuse of narcotics and alcohol independence 10) Allergy to experimental drug and other contraindication 11) Advanced tumor patients 12) Neuromuscular blockade other than for intubation 13) Pregnancy or lactation 14) Patient that participate other trial at past 30 days -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Ventilation duration | From intubation to weaning from mechanical ventilation, up to 7 days.
  The time of intubation and the time of weaning from mechanical ventilation are recorded.

SECONDARY OUTCOMES:
Delirium | From the beginning of sedation to discharge from ICU, up to 28 days.
  Using the Mini-mental State Examination(MMSE) to examine the delirium.
Blood pressure | From the beginning to weaning of sedation, up to 7 days.
  blood pressure is recorded.
Cost of sedation drug | From the admition to discharge from ICU,up to 28 days.
  The cost of sedation drug is calculated.
Cost of narcotics | From the admition to discharge from ICU,up to 28 days.
  Cost of narcotics is calculated.
Cost of ICU stay | From the beginning to weaning of sedation, up to 7 days.
Heart rate | From the beginning to weaning of sedation, up to 7 days.
Respiration Rate | From the beginning to weaning of sedation, up to 7 days.
Pulse blood oxygen saturation | From the beginning to weaning of sedation, up to 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, Professor, Principal Investigator — Tianjin Third Central Hospital